CLINICAL TRIAL: NCT05298176
Title: Combining Afatinib and Concurrent Chemotherapy, Followed by Osimertinib and Concurrent Chemotherapy, in Untreated EGFR Positive NSCLC Tumors
Acronym: COMBINATION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Idris Bahce, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL74383.029.20; 2020-003025-37 (EudraCT Number)
Record Dates: First submitted 2022-01-15; First posted 2022-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: EGFR; EGFR mutation; Afatinib; Osimertinib; Chemotherapy; Combination strategy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib; osimertinib; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with untreated EGFR positive NSCLC tumors (Experimental): TKI-naïve advanced NSCLC patients, harboring a non-exon20insertion uncommon EGFR mutation, who are eligible for treatment with afatinib in 1st line
  Interventions: Drug: Afatinib, Osimertinib, Carboplatin and Pemetrexed

INTERVENTIONS:
Drug: Afatinib, Osimertinib, Carboplatin and Pemetrexed — This study consists of 2 parts. Part 1 is defined as a first line treatment with afatinib orally (30 mg once a day) for the first 6 weeks, followed by concurrent use of afatinib (20mg once a day, part 1B) plus 2 cycles of carboplatin and pemetrexed (21 days per cycle); followed by afatinib monotherapy (30mg once a day). Part 2 comprises a 2nd line treatment with osimertinib (80 mg once daily) after failure of part 1, only in T790M positive patients for the first 6 weeks, followed by concurrent use of osimertinib (80mg once a day) plus 2 cycles of carboplatin and pemetrexed (21 days per cycle); followed by osimertinib monotherapy (80mg once a day).

SUMMARY:
The aim of the COMBINATION trial is to prospectively study the sequential approach of using afatinib combined with a short course of chemotherapy, followed by osimertinib, upon progression and acquisition of a T790M mutation, also combined with a short course of chemotherapy.

DETAILED DESCRIPTION:
The investigators hypothesized that treating advanced stage EGFR mutation positive NSCLC in first line with afatinib and osimertinib in second line (in T790M positive tumors) will cause an apoptotic cell death in a large part of TKI-sensitive cancer cells, resulting in a large reduction of the tumor bulk. Adding cytotoxic chemotherapy after 6 weeks of EGFR-TKI will destroy remaining TKI-resistant subclones at an early stage, when the TKI-resistance tumor volume is the smallest and most vulnerable. The investigators will administer only 2 cycles of chemotherapy to limit toxicity, while maintaining a substantial anti-cancer effect. After progression on afatinib-chemotherapy combination, some participants will develop T790M and will be able treated by osimertinib-chemotherapy combination.

So, this strategy will allow the investigators to timely sequence the most appropriate drugs (afatinib and osimertinib with chemotherapy) to get the highest anti-cancer efficiency. In this way, the investigators will avoid long periods of maintenance treatments with chemotherapy or anti-VEGFR treatments that are associated with toxicity, costs, and necessitate the participants to come into the ward for intravenous medication. The limited cycles of chemotherapy also allows the treating physician to again treat the participant with the same chemotherapy regimen once progression occurs after all sensible targeted therapy options have been used.

Therefore, the investigators hypothesize that this sequential combination strategy will be more effective than other available strategies and will improve the quality of patient care as compared to current general practice.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed NSCLC, positive for non-exon20insertion uncommon EGFR mutations that are eligible for afatinib therapy in first line
2. WHO PS 0-2
3. Be willing and able to provide written informed consent for the trial.
4. Be above 18 years of age on day of signing informed consent.
5. Patients must have radiological measurable disease
6. Demonstrate adequate organ function, as deemed acceptable by the treating physician in the context of metastatic NSCLC.

Exclusion Criteria:

1. Inability to provide informed consent
2. Inability to take study medications
3. Patients with symptomatic or unstable CNS metastases
4. Prior EGFR TKI or platinum-doublet therapy for advanced stage NSCLC. Prior (neo)adjuvant treatments are allowed when the last administration is one year or more.
5. Evidence of interstitial lung disease or active, non-infectious pneumonitis.
6. Active infection requiring systemic therapy.
7. Active Hepatitis B or C.
8. Psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
9. Patient is pregnant or breastfeeding, or expecting to conceive within the projected duration of the trial, starting with the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Disease control rate (DCR) | 18 months
  To assess the efficacy of the sequential strategy of front-line afatinib-chemo, followed by a treatment with osimertinib-chemo in those patients that develop a T790M mutation as a mechanism of resistance

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From start of therapy until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 50 months
  To assess long term efficacy
Overall Survival (OS) | From start of therapy until the date of death from any cause, assessed up to 50 months
  To assess long term efficacy
Objective response rate according to RECIST v1.1 after start of afatinib | At 6 weeks
  To assess short term efficacy
Objective response rate according to RECIST v1.1 after start of afatinib | At 12 weeks
  To assess short term efficacy
Objective response rate according to RECIST v1.1 after start of osimertinib | At 6 weeks
  To assess short term efficacy
Objective response rate according to RECIST v1.1 after start of osimertinib | At 12 weeks
  To assess short term efficacy
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From start of therapy until disease progression or study drug toxicity assessed up to 100 days after part 1 and 2
  To assess the safety of afatinib and osimertinib intercalated with 2 cycles of carboplatin-pemetrexed

CONTACTS AND LOCATIONS:
Overall Officials: Idris Bahce, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam UMC, location VUmc, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided